CLINICAL TRIAL: NCT04702607
Title: Pilot Study to Assess Lung Function Using Perfusion Blood Volume Dual Energy CT and 4DCT Derived Lung Ventilation Imaging
Brief Title: Functional Lung Imaging With DECT and 4DCT
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 18520
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- contrast enhanced 4DCT
  Interventions: Procedure: contrast enhanced 4DCT

INTERVENTIONS:
Procedure: contrast enhanced 4DCT — Functional Lung Imaging with DECT and 4DCT

SUMMARY:
The basic premise of this pilot study is to enroll 40 patients over 3 years who have Stage II, III, or IV non-small cell lung cancer and are planned for definitive treatment with concurrent chemoradiation where a contrast enhanced 4DCT is planned.

ELIGIBILITY:
Inclusion criteria:

* Patients have histologic diagnosis of non-small cell lung cancer
* Patients have AJCC stage II, III or IV disease were the plan is to receive definitive concurrent chemoradiation to 60 Gy or higher
* Age > 18 years of age
* Patients are able to provide informed consent
* No additional lung radiation is planned until after the 2nd CT on this study (i.e. patient does not have a solitary pulmonary nodule or second primary that the plan is to undergo SBRT)
* Patient must have adequate kidney function to receive IV contrast (following institutional policy supplied by radiology). The cutoff level for serum creatinine is 1.6 mg/dL
* Negative urine pregnancy test before every CT scan

Exclusion criteria:

* Allergy to IV iodine contrast
* Severe claustrophobia
* Further thoracic radiation therapy is planned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients have histologic diagnosis of non-small cell lung cancer
  * Patients have AJCC stage II, III or IV disease were the plan is to receive definitive concurrent chemoradiation to 60 Gy or higher
  * Age > 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2024-10-05 (Actual)

PRIMARY OUTCOMES:
evaluate the reproducibility of PBV DECT imaging and 4DCT derived lung ventilation for evaluating lung function | 3 years
correlate changes of PBV DECT and 4DCT lung function images seen at ~6 months with radiation dose and with patient reported outcome quality of life | 3 years

SECONDARY OUTCOMES:
• To propose a novel biologic (i.e. functional) dose volume algorithm to reduce PBV and 4DCT lung function changes | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Feigenberg, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abamson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No